CLINICAL TRIAL: NCT03449732
Title: Evaluation of the Pupil Dilation Reflex (PDR) Using a Pupillary Pain Index (PPI) Stimulation Protocol in Response to Noxious Stimulation in Anaesthetized Children. A Proof of Concept Trial
Brief Title: Evaluation of the Pupil Dilation Reflex in Response to Noxious Stimulation in Anaesthetized Children. A Proof of Concept Trial
Acronym: Pain@OR-kids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Davina Wildemeersch, Principle investigator, University Hospital, Antwerp
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 17/46/519
Record Dates: First submitted 2018-02-22; First posted 2018-02-28 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Pain; Monitoring, Intraoperative
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PDR measurement group A (Experimental): Two measurements of PDR perioperatively before and after opioid administration in toddlers (28 days until 23 months)
  Interventions: Device: PDR measurement
- PDR measurement group B (Experimental): Two measurements of PDR perioperatively before and after opioid administration in children (2 until 11 years)
  Interventions: Device: PDR measurement
- PDR measurement group C (Experimental): Two measurements of PDR perioperatively before and after opioid administration in adolescents (12 until 18 years)
  Interventions: Device: PDR measurement

INTERVENTIONS:
Device: PDR measurement — PDR measurement at two standardized times perioperatively:
  1. Anesthetized subject by sevoflurane sedation until a minimum alveolar concentration (MAC) of at least 1,5 is reached
  2. Administration of fentanyl 2µg/kg, in the absence of adjustments in sedation depth
  Other Names: PPI assessment

SUMMARY:
After conduction a pilot study, pupillary dilation reflex (PDR) is measured in response to nociceptive stimulation perioperatively in infants, children and adolescents.

DETAILED DESCRIPTION:
An infrared camera of the video pupillometer measures the pupillary dilation reflex (PDR) in response to incremental nociceptive stimuli. The PDR is a robust reflex, even in patients under general anesthesia, and may provide a potential evaluation of the autonomous nociceptive circuit. American Society of Anesthesiologists (ASA) classification I or II patients from the age of 28 days till 18 years undergoing elective surgery under general anesthesia are recruited. Enrolled patients perioperative undergo PDR measurement at 2 different standardized times (before and after opioid administration) generated by an inbuilt pupillary pain index (PPI) protocol. PPI, as a surrogate for nociception includes noxious stimulations from 10 up to 60 milli ampere (mA) until pupil dilation is larger than 13% from baseline diameter. Therefore, no inappropriate high stimulation is executed.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled abdominal, urological or otorhinolaryngology surgery under general anaesthesia
* ASA I-II

Exclusion Criteria:

* History of eye deformity, invasive ophthalmologic surgery
* Known cranial nerve(s) deficit
* Infection of the eye
* Predicted difficult airway management (Paediatric Difficult Airway Guidelines - Difficult Airway Society)
* Chronic opioid use (>3 months)
* Ongoing treatment with beta-blockers, dopamine antagonists, topical atropine
* Preoperatively administrated benzodiazepins or antiemetics

Ages: 28 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2018-03-30 (Actual); Primary Completion 2021-04-26 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Stimulation Intensity | During pupil measurements in the perioperative period
  Necessary stimulation intensity to dilate the pupil more than 13%

SECONDARY OUTCOMES:
Pupillary Pain Index score | During pupil measurements in the perioperative period
  Device specific PPI score defined in accordance to stimulation intensity necessary for pupil dilation more than 13%
Blood pressure | During PDR measurements
  Hypertension as a common used parameter for perioperative nociceptive assessment defined as an increase in systolic blood pressure by >10% of the initial systolic blood pressure
Heart rate | During PDR measurements
  Tachycardia as a common used parameter for perioperative nociceptive assessment

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Kegels, MD, Principal Investigator — University Hospital, Antwerp; Vera Saldien, MD, Study Chair — University Hospital, Antwerp
Locations (1):
- University hospital Antwerp, Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: Undecided